CLINICAL TRIAL: NCT01617343
Title: The HEP-OKS Pilot Study - a Randomized Controlled Trial of Hemifield Eye Patching and Optokinetic Stimulation to Treat Hemispatial Neglect in Stroke Patients
Brief Title: The HEP-OKS Study - Hemifield Eye Patching and Optokinetic Stimulation to Treat Hemispatial Neglect in Stroke Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Luebeck (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Bjoern Machner, MD, Principal Investigator, University of Luebeck
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HEP-OKS-01
Record Dates: First submitted 2012-06-05; First posted 2012-06-12 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Spatial Neglect; Cerebral Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention): Patients in this control group will receive usual care following stroke including standard physiotherapy and occupational therapy.
- HEP-OKS (Experimental)
  Interventions: Behavioral: hemifield eye patching (HEP) + optokinetic stimulation (OKS)

INTERVENTIONS:
Behavioral: hemifield eye patching (HEP) + optokinetic stimulation (OKS) — Patients in this arm will wear standard spectacle frames containing noncorrective lenses to which right half-field patches are attached (hemifield eye patching, HEP). In case of patients already wearing prescribed glasses, the patches will be attached to their own glasses. The glasses will be worn all-day for the duration of the treatment phase (seven days) and only be removed for sleeping and face cleaning as well as for the duration of the daily OKS treatment sessions.
  Furthermore these patients will receive daily sessions (20 minutes) of optokinetic stimulation (OKS). Therefore patients will be seated in front of a widescreen monitor, watching a black background with a pattern of various objects (size 1°), which coherently and continuously move to the left at a velocity of 10 °/s.
  Arms: HEP-OKS

SUMMARY:
Spatial neglect represents one of the major cognitive disorders following stroke. Patients patients fail to be aware of objects or people to their left and orientate instead to their right side. Enduring neglect has been found to be a poor prognostic indicator for functional independence following stroke. Despite some promising experimental accounts there are no established treatments for this condition.

The aim of this study is to test whether a combined treatment with hemifield eye patching (HEP) and optokinetic stimulation (OKS) can permanently reduce neglect behaviour and improve functional outcome in patients with hemispatial neglect following stroke.

The investigators hypothesise that the treatment with HEP and OKS will lead to a greater reduction of neglect scoring in the neglect test battery as well as a greater improvement in functional independence scores as compared to the spontaneous clinical course of the usual-care control group.

DETAILED DESCRIPTION:
To specify, this study should answer the following main question: Does the daily wearing of hemifield eye patches over a period of 1 week in combination with daily sessions of optokinetic stimulation lead to a significant reduction of neglect behaviour as measured by total scores in a paper-and-pencil neglect test battery and/or an improvement in functional independence scores (Catherine-Bergego-Scale, Barthel Index) in a cohort of stroke patients with acute hemispatial neglect as compared to the spontaneous course of the disease in a control patient group without a neglect-specific treatment?

ELIGIBILITY:
Inclusion Criteria:

* Right hemisphere stroke
* Spatial neglect as determined by pathological scores in at least two tests of a neglect test battery (Azouvi et al., JNNP, 2004)
* Age > 18 years old
* Informed consent signature

Exclusion Criteria:

* Bilateral or previous unilateral stroke lesions
* Pre-existing neurodegenerative disease
* Inability to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Total score in a neglect test battery | Change from baseline at Day 8 (post-treatment)
  Performance in a neglect test battery (score between 0 and 100%) consisting of standard neglect tests including two cancellation tasks, line bisection, figure copying and text reading
Functional independence score | Change from baseline at Day 8 (post-treatment)
  Level of functional independence (score between 0 and 100%) as measured by the Barthel-Index and the Catherine-Bergego-Scale

SECONDARY OUTCOMES:
Performance in paper-and-pencil subtests | Change from baseline at Day 8 and at Day 30
  The secondary outcome measures include scores of the individual subtests of the neglect test battery, i.e. bells and star cancellation tasks, line bisection, figure copying and text reading.
Performance in computerized attention tests | Change from baseline at Day 8 and at Day 30
  Performance in two computerized attention tests. These comprise a Posner Attention Task and a visual search task including eye movement analyses.
MRI | Day 1
  All patients (without contraindications) undergo cranial Magnetic Resonance Imaging (MRI) including 3D lesion analysis, resting state fMRI and a task-related fMRI with optokinetic stimuli. Patients' MRI data will be correlated to behavioural performance (see primary and other secondary outcome measures) and will also be compared to controls without spatial neglect.
Total score in the neglect test battery at follow-up | Change from baseline at Day 30
  For details please see primary outcome measure
Functional independence score at follow-up | Change from baseline at Day 30
  For details please see primary outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Bjoern Machner, MD, Principal Investigator — University of Luebeck
Locations (1):
- University of Luebeck, Dept. of Neurology, Lübeck, Schleswig-Holstein, Germany

REFERENCES:
- [Derived] Machner B, Konemund I, Sprenger A, von der Gablentz J, Helmchen C. Randomized controlled trial on hemifield eye patching and optokinetic stimulation in acute spatial neglect. Stroke. 2014 Aug;45(8):2465-8. doi: 10.1161/STROKEAHA.114.006059. Epub 2014 Jun 12. PMID 24923723